CLINICAL TRIAL: NCT00420290
Title: Inflammation, Proteolysis and IL-1 Beta Receptor Inhibition in Chronic Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Adriana Hung, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060661
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Results first posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-10

CONDITIONS: End Stage Renal Disease
Keywords: inflammation; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kineret (Active Comparator): Interleukin-1 receptor antagonist
  Interventions: Drug: kineret
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: kineret — 100 mg administered subcutaneously every other day (3 days a week during hemodialysis) for 4 weeks
  Other Names: Anakinra
  Arms: Kineret
Drug: placebo — 100 mg administered subcutaneously every other day (3 days a week during hemodialysis) for 4 weeks
  Arms: Placebo

SUMMARY:
Chronic hemodialysis (CHD) patients display multiple metabolic abnormalities related to advanced uremia. Despite vigorous attempts to prevent these abnormalities and their consequences, most CHD patients suffer from a unique form of nutritional derangement, which can be termed as "uremic wasting". Several studies have demonstrated that the presence of uremic wasting, especially the degree of loss of muscle mass, sharply increases mortality and hospitalization rate in CHD patients.

Several factors have been thought to be associated with uremic wasting, including hormonal derangement, anorexia, physical inactivity, and concurrent illnesses. Chronic inflammation, also highly prevalent in these patients, causes muscle catabolism in animal models and certain clinical conditions. Epidemiological studies show an association between chronic inflammation and uremic wasting in hemodialysis patients indicating a possible causal relationship.

The cause for the activated inflammatory state in CHD patients is believed to be multi-factorial. Nevertheless, it is certainly important for the host to limit its biological activity by eliciting a stronger anti-inflammatory response, for example through the production of naturally occurring receptor antagonist. Interleukin 1 beta, one of the major pro-inflammatory cytokines has been shown to be associated with protein catabolism in several chronic disease states, including advanced uremia. A balance between interleukin 1 beta (agonist) and its naturally occurring receptor antagonist IL-1ra may play a pivotal role in controlling the inflammatory response and its consequences in this population.

The overall goal of this particular grant application is to examine the short-term effects of the administration of the recombinant form of IL-1ra on 1) chronic inflammatory state and 2) protein homeostasis in chronically inflamed CHD patients.

We have updated our protocol to perform an interim analysis. The interim analysis will be performed after half of the planned study sample has been enrolled (14 subjects; 7 in each arm). The interim analysis has been approved by the Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on CHD for more than 3 months;
2. Ability to read and sign the consent form;
3. Have acceptable dialysis adequacy (Kt/V > 1.2);
4. Use biocompatible hemodialysis membrane;
5. Have a patent, well functioning, arteriovenous dialysis access;
6. Signs of chronic inflammation (the average of three consecutive CRP measurements ≥ 5 mg/L).

Exclusion Criteria:

1. Patients with residual renal function > 5 ml/min or urine output > 100 ml/day;
2. Pregnancy;
3. Intolerance to the study medication or contraindication to the study medication: Hypersensitivity to E. coli-derived proteins, anakinra, or any component of the formulation; patients with active infections (including chronic or local infection);
4. Severe, unstable, active, or chronic inflammatory disease (active infection, active connective tissue disorder, active cancer or cancer history in the prior 5 years, HIV, liver disease including positive test or history of Hepatitis B or C);
5. Hospitalization within 1 month prior to the study;
6. Malfunctioning arterial-venous vascular access [recirculation and/or blood flow < 500 ml/min for an arterial-venous graft (AVG) or < 400 ml/min for an arterial-venous fistula (AVF)];
7. Patients receiving steroids and/or other immunosuppressive agents;
8. Life-expectancy less than 6 months;
9. Age greater than 75 or less than 18 years old;
10. Hypersensitivity to organic nitrates, isosorbide, or nitroglycerin.
11. Presence of active infections or a history of pulmonary TB infection with or without documented adequate therapy. Subjects with current active TB, or recent close exposure to an individual with active TB, are excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Hung, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Hung AM, Ellis CD, Shintani A, Booker C, Ikizler TA. IL-1beta receptor antagonist reduces inflammation in hemodialysis patients. J Am Soc Nephrol. 2011 Mar;22(3):437-42. doi: 10.1681/ASN.2010070760. Epub 2011 Feb 10. PMID 21310819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Vanderbilt University Medical Center and Nashville Veterans Affairs Outpatient Dialysis units between January 2008 and May 2010.
Pre-assignment Details: There is a 3-month screening period following enrollment to determine level of inflammation. To be eligible to participate in the intervention phase of the study and be assigned to a group, participants must have three consecutive CRP levels > 5 mg/L. Although 31 subjects were enrolled, only 22 were eligible to be assigned to a group.
Groups:
- Kineret: 100 mg Interleukin-1 receptor antagonist administered subcutaneously every other day (3 days a week during hemodialysis) for 4 weeks
- Placebo: 100 mg placebo administered subcutaneously every other day (3 days a week during hemodialysis) for 4 weeks
Period: Overall Study
Arm/Group | Kineret | Placebo
Started | 11 | 11
Completed | 7 | 7
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — did not meet inclusion/exclusion | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kineret | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (10.5) | 50 (11.4) | 47 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: High Sensitivity C-reactive Protein (hsCRP)
Description: hsCRP is a sensitive laboratory assay for serum levels of C-reactive protein, which is a biomarker of inflammation.
Time Frame: month 1
Population: The number of participants for analysis was based on those subjects who completed the 4-week study. The analysis was per protocol.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Kineret | Placebo
Number analyzed (Participants) | 7 | 7
mg/dl | 4.67 (2.87) | 15.11 (10.18)
Statistical Analysis 1: Comparison: Kineret vs Placebo; Using data from 128 CHD patients, CRP data were highly skewed, and data were log transformed to achieve normality. With 14 pts in each group (total of 28), it was predicted the minimum detectable difference between control and intervention would be 15% (1.22 for control group and 1.00 for the intervention group), with an 80% power and an alpha of 0.05 using t test approach. Thus, planned sample size was 30 to complete the study; Test type: Superiority or Other; p = 0.008, ANCOVA — 0.031 is the upper level of significance

2. Secondary Outcome: Interleukin-6 (IL-6)
Description: IL-6 is a sensitive laboratory assay for serum levels of interlukin-6, which is a pro-inflammatory cytokine that is used to evaluate the inflammatory response.
Time Frame: month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Kineret | Placebo
Number analyzed (Participants) | 7 | 7
pg/ml | 3.34 (3.09) | 8.14 (6.04)
Statistical Analysis 1: Comparison: Kineret vs Placebo; Test type: Superiority or Other; p = 0.03, ANCOVA

3. Secondary Outcome: Serum Prealbumin
Description: Prealbumin is a sensitive laboratory assay for serum levels of prealbumin, which is a biomarker of nutrition.
Time Frame: month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Kineret | Placebo
Number analyzed (Participants) | 7 | 7
mg/dl | 46.43 (11.27) | 33.57 (12.23)
Statistical Analysis 1: Comparison: Kineret vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

4. Secondary Outcome: Serum Albumin
Description: Albumin is a sensitive laboratory assay for serum levels of albumin, which is a biomarker of nutrition.
Time Frame: month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Kineret | Placebo
Number analyzed (Participants) | 7 | 7
g/dl | 4.26 (0.40) | 3.95 (0.38)
Statistical Analysis 1: Comparison: Kineret vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

5. Secondary Outcome: Lean Body Mass (LBM)
Description: LBM is a measurement of body composition in terms of lean body mass as determined using Dual Energy X-ray Absorptiometry (DEXA) performed 1 to 2 hours after dialysis.
Time Frame: month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Kineret | Placebo
Number analyzed (Participants) | 7 | 7
kg | 59.13 (8.72) | 50.38 (7.86)
Statistical Analysis 1: Comparison: Kineret vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Kineret | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kineret (N=7) | Placebo (N=7)
injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
hemodialysis access site infection (Infections and infestations) | 1 (1) | 0 (0)
injection site hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 1 (1) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size is small and the intervention is of short duration. Also, the results cannot be generalized to all CHD patients because our inclusion criteria were stringent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes